CLINICAL TRIAL: NCT03127033
Title: Patient Satisfaction of Soft Liner Versus Acrylic Resin Telescopes in Complete Overdenture Patients With Ectodermal Dysplasia: Non-Randomized Clinical Trial
Brief Title: Comparison Between Acrylic and Soft Liner Telescopic Overdentures Regarding Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Hisham Abd El rahman Mohsen, Principal investigator, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 171088
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Patient Satisfaction; Retention; Periodontal Health
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Soft liner telescopes — Soft liner telescopes: Overdenture will be adjusted by relieving acrylic opposite to the abutment about 2 mm using a metal stone. The relieved areas will be painted with an adhesive and the rest of the fitting surface of the denture will be painted with a separating medium.
  The soft liner (Silicone based soft liner, mollosil, chairside soft relining-long term, DETAX, Germany) will then be applied in the relieved areas to act as a secondary coping The base and catalyst will be mixed according to the manufacturer's instructions on a glass slab. The mix will be placed on the relieved area, seated in the patient's mouth, the patient is asked to bite in centric relation and the excess liner is removed with a lancet.

SUMMARY:
Conventional complete overdenture will be made to ectodermal dysplasia patients, a week after delivery and after 3 months Patient satisfaction, retention and periodontal condition will be assessed. the denture will be taken from the patient for 2 weeks.Acrylic telescopes will be replaced with soft liner and again Patient satisfaction, retention and periodontal condition will be assessed a week after delivery and 3 months later.

DETAILED DESCRIPTION:
Upper and Lower Primary impressions will be carried out by using irreversible hydrocolloid (Alginate, Tropicalgin, Normal setting, Zhermack, Italy) according to manufacturer's instructions using stainless steel stock trays.

Secondary upper impression is done with an acrylic special tray. Border molding is done with putty consistency rubber base impression material, Final impression with medium consistency rubber-base impression material (Silicone impression material, Elite P&P, Regular Body-Normal set, Zhermack, Italy) Maxilla-mandibular relationship will be recorded using check bite technique. Setting of artificial teeth will be performed and trial dentures will be tried in inside patients' mouth.

The finished and polished dentures will be delivered immediately after the necessary occlusal adjustments and instructions regarding hygiene and maintenance.

The patient will use the upper overdenture for 3 months. The overdenture is taken from the patient for two weeks, after which the maxillary overdenture will be adjusted by relieving acrylic opposite to the abutment about 2 mm using a metal stone. The relieved areas will be painted with an adhesive and the rest of the fitting surface of the denture will be painted with a separating medium.

The soft liner (Silicone based soft liner, mollosil, chairside soft relining-long term, DETAX, Germany) will then be applied in the relieved areas to act as a secondary coping The base and catalyst will be mixed according to the manufacturer's instructions on a glass slab. The mix will be placed on the relieved area, seated in the patient's mouth, the patient is asked to bite in centric relation and the excess liner is removed with a lancet.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous ectodermal dysplasia patients with few remaining teeth.
2. Cooperative patients with no history of psychological diseases.
3. Length of maxillary remaining teeth should not be less than 4mm.

Exclusion Criteria:

- 1- Patients with tempo-mandibular joint disorders or systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.

2- Patients allergic to acrylic resin.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 3 months
  A questionaire will be given to the patient to assess thier denture satisfaction in numerical data using Visual Analogue Scale

SECONDARY OUTCOMES:
Retention | 3 months
  Retention will be assessed subjectively using Kapur's retention scoring system in ordinal data.
Gingival index | 3 months
  periodontium condition will be assessed through Gingival index scoring system in ordinal data
Probing depth | 3 months
  Probing depth will be measured using periodontal probe in Mm
Tooth mobility | 3 months
  tooth mobility will be assessed through periostest using Periotest value.
Absence or presence of inflammation | 3 months
  Absence or presence of inflammation will be assessed visually as a binary outcome

IPD SHARING:
Plan to Share IPD: No